CLINICAL TRIAL: NCT04295447
Title: A Randomized, Open-label, Phase 2 Study of Adjuvant Apalutamide or Standard of Care in Subjects With High-risk, Localized or Locally Advanced Prostate Cancer After Radical Prostatectomy
Brief Title: Adjuvant Apalutamide in Subjects With High-risk Localized or Locally Advanced Prostate Cancer After Radical Prostatectomy
Acronym: ADAM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universität Münster (Other)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKM17_0018
Record Dates: First submitted 2020-02-20; First posted 2020-03-04 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Prostatic Neoplasms
Keywords: prostate cancer; apalutamide; radical prostatectomy; randomized; high risk adenocarcinoma; neoplasm
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Standard of Care; apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Other): 1. Observation only or
  2. An optional adjuvant radiation of the prostate bed in case of positive surgical margin
  Interventions: Other: Standard of care
- Apalutamide (Experimental): 30 cycles apalutamide 240 mg (4 x 60 mg) once daily on days 1-28 of a 28-day cycle in addition to standard of care
  Interventions: Other: Standard of care; Drug: Apalutamide 60Mg Tab

INTERVENTIONS:
Other: Standard of care — 1. Observation only or
  2. An optional adjuvant radiation of the prostate bed in case of positive surgical margin
Drug: Apalutamide 60Mg Tab — (4 x 60 mg) once daily on days 1-28 of a 28-day cycle
  Arms: Apalutamide

SUMMARY:
The primary objective of this trial is to determine if adjuvant apalutamide in prostate cancer patients at high risk of developing subsequent metastatic disease results in prolonged biochemically recurrence-free survival after radical prostatectomy (RPE) in comparison to standard of care (SOC).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF).
2. Men ≥ 18 years of age.
3. Patients with histologically confirmed adenocarcinoma of the prostate after radical prostatectomy.
4. Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1.
5. Exclusion of metastatic disease by computed tomography (CT)-scan of abdomen (magnetic resonance imaging (MRI) of abdomen is possible) and bone scan prior to study inclusion. A PSMA PET-CT/MRI is possible. In this case it has to be done with a diagnostic CT/MRI with contrast media and not with a low dose CT-scan only. In case PSMA-PET imaging has been done, a bone scan can be omitted. CT/MRI, and bone-scan imaging or PSMA PET-CT/MRI administered ≤12 weeks before RPE may be used for screening.
6. Patients after radical prostatectomy must meet the d'Amico criteria for high risk of disease recurrence: i.e. one of the following after RPE: 1) Gleason score ≥8, any T-stage, any initial PSA (iPSA) or 2) Gleason score 6 or 7, any iPSA and ≥pT3c or 3) iPSA >20 ng/ml, any Gleason score, any T-stage.
7. Patients have to have recovered from radical prostatectomy within four weeks to be able to take part in the study.
8. PSA-value must have declined below 0.2 ng/ml prior to randomization
9. Adequate hematologic, hepatic, and renal function:

   Hematologic
   * Haemoglobin ≥9.0 g/dL independent of transfusions
   * Neutrophils ≥1.5 Ths./µL

   Hepatic:
   * Total bilirubin ≤1.5X upper limit of normal (ULN) [except for subjects with documented Gilbert's disease in which case total bilirubin not to exceed 10X ULN]
   * Alanine (ALT) and aspartate (AST) aminotransferase ≤2.5X ULN

   Renal:
   * Serum creatinine <1.5X ULN or calculated creatinine clearance ≥50 mL/min
   * Serum potassium ≥3.5 mM
   * Serum albumin ≥ 3.0 g/dL.
10. Ability to swallow study medication tablets.
11. In case of apalutamide treatment: Agrees to use a condom and another highly effective method of birth control if he is having sex with a woman of childbearing potential or to use a condom if he is having sex with a woman who is pregnant

Exclusion Criteria:

1. Any chronic medical condition requiring a higher dose of corticosteroid than 10mg prednisone/prednisolone q.d.
2. Prior cytotoxic chemotherapy or biologic therapy for the treatment of prostate Cancer.
3. Prior or current treatment of prostate cancer with apalutamide, enzalutamide, darolutamide, or other investigational agents targeting the androgen receptor.
4. Prior therapy with Sipuleucel-T or other vaccination or immunogenic therapy for the treatment of prostate Cancer.
5. Prior treatment with abiraterone acetate or other androgen synthesis inhibitors (e. g. ketoconazole, TAK700, TOK001).
6. Use of 5-α reductase inhibitors (eg, dutasteride, finasteride) ≤4 weeks prior to randomization.
7. Prior surgical castration or medical castration using LHRH-Agonists or GnRH-Antagonists.
8. Prior or current radiation or radionuclide (including radium-223 dichloride) therapy for treatment of prostate cancer (adjuvant radiation of the prostate bed without involvement of the regional lymph node template as by standard of care in case of positive surgical margins (R1) is allowed).
9. Prior or current systemic treatment with an azole drug (e.g. fluconazole, itraconazole) within 4 weeks of Cycle 1, Day 1.
10. Any lymph node or distant metastasis.
11. History of seizure or condition that may predispose to seizure (including, but not limited to prior stroke, transient ischemic attack or loss of consciousness ≤1 year prior to randomization; brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect).
12. Current or prior treatment with anti-epileptic medications for the treatment of seizures.
13. Management of cardiovascular risk factors, such as hypertension, diabetes or dyslipidaemia should be optimised as per standard of care before treatment with apalutamide will be initiated

    13.1. Uncontrolled hypertension (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg. For patients with relevant comorbidities (e.g. diabetes) systolic BP ≥130 mmHg or diastolic BP ≥80 mmHg). Patients with a history of hypertension are allowed provided that blood pressure is controlled by anti-hypertensive Treatment

    13.2. Patients with uncontrolled diabetes defined as HbA1c ≥7.5%

    13.3. Patients with a dyslipidemia defined as LDL cholesterol >100 mg/dl. For patients with a dyslipidemia defined as LDL cholesterol >100 mg/dl and SCORE-value of 1-5%: In case of a SCORE-value of <1% a LDL cholesterol level of up to 115 mg/dl is acceptable. In case of increased LDL cholesterol above these values a statin-therapy can be initiated and a rescreening within 4 weeks is possible

    13.4. Cardiovascular risk assessment via an appropriate score (e.g. the SCORE-Chart for the European high/low risk score from the European Society of Cardiology) and ≥ borderline risk i.e. 10% of developing cardiovascular events within 10 years without prior established cardiovascular disease
14. Active or symptomatic viral hepatitis or chronic liver disease or HIV.
15. History of pituitary or adrenal dysfunction.
16. Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of <50% at baseline.
17. Any condition that requires treatment with digoxin, digitoxin, and other digitalis drugs.
18. Long QT-Syndrome.
19. Atrial Fibrillation, or other cardiac arrhythmia requiring therapy.
20. Other malignancy with a ≥30% probability of recurrence within 24 months, except non-melanoma skin Cancer.
21. Any condition, which, in the opinion of the investigator, would preclude participation in this trial.
22. Gastrointestinal conditions affecting Absorption.
23. Hypersensitivity to the active substance, or to any of the excipients of the study medication.
24. Any psychological, cognitive, familial, sociological or geographical condition that, in the investigator's opinion, compromises the patient's ability to understand the patient information, to give informed consent or to comply with the study protocol.
25. Participation in another interventional clinical trial during this trial or within 4 weeks before entry into this trial. There may be exceptions at the discretion of the (coordinating) investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS). | From date of randomization until the date of first documented progression (BCR or metastases) or date of death from any cause, whichever came first, assessed up to 7 years"
  This endpoint is defined as time interval from randomization until BCR (irrespective of the PSADT), metastases, or death from any cause, whichever occurs first. BCR is defined as a PSA ≥ 0.2 ng/ml that has risen on at least two separate occasions at least four weeks ± 3 days apart and measured by the central PSA-lab. The time of BCR is then backdated to the time of the first increased PSA measurement.
  Metastatic disease will be defined as the presence of bone metastases visualized on bone scan prostate cancer working group 3 (PCWG3)-criteria; and/or visceral (e.g. liver, lung, brain) or extra-pelvic nodal metastases visualized on CT scan (or MRI scan) (RECIST 1.1-criteria). Evaluations will be performed every 6 months once BCR occurred or sooner if clinically indicated.
  For a patient with none of these events before the end of follow-up, observation of PFS will be censored at the date of his date of last contact.

SECONDARY OUTCOMES:
PSA doubling time (PSADT) | If BCR occurs up to 6 months later
  In case of a BCR, PSA kinetics as the PSADT are calculated based on the monthly PSA measurements during the first six months after the BCR. The values used to determine the BCR are included in the calculation of PSA kinetics as well.
  PSADT is calculated according to Pound et al. by the natural log of 2 (0.693) divided by the slope of the relationship between the log of PSA and time of PSA measurement (i.e. time from BCR) for each patient [33]. PSADT can also be assessed using the MSKCC PSADT calculator (https://www.mskcc.org/nomograms/prostate/psa_doubling_time) using the above definitions.
Incidence of Adverse Events [Safety and Tolerability] | From date the informed consent is signed until BCR occured and PSADT was calculated or when distant metastasis occurred (both with or without BCR) or date of death from any cause, whichever came first, assessed up to 7 years.
  Safety and tolerability assessed on the basis of adverse events, more precisely adverse events, serious adverse events, adverse reactions, and serious adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bögemann, Univ.-Prof. Dr. med., Principal Investigator — Universitätsklinikum Münster, Klinik für Urologie und Kinderurologie
Locations (21):
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Uniklinikum Salzburg, Landeskrankenhaus, Salzburg
  - Hanusch-Krankenhaus, Vienna
- Germany (17):
  - University Hospital Münster, Münster, North Rhine-Westfalia
  - Universitätsklinikum Augsburg Klinik für Urologie, Augsburg
  - GFO Kliniken Rhein-Berg, Bergisch Gladbach
  - Urologische Partnerschaft Köln, Cologne
  - Urologicum Duisburg, Duisburg
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - St. Antonius-Hospital Gronau GmbH Klinik für Urologie, Kinderurologie und Urologische Onkologie, Gronau
  - Universitätsklinikum Jena, Jena
  - KLINIKUM LANDSHUT gemeinnützige GmbH, Landshut
  - Klinikum Leverkusen gGmbH, Klinik für Urologie, Leverkusen
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinikum Magdeburg, Magdeburg
  - Klinik für Urologie, Lehrstuhl Regensburg, Am Caritas Krankenhaus St. Josef, Regensburg
  - UroGynZentrum, Wuppertal
  - Helios Universitätsklinikum Wuppertal, Universität Witten/Herdecke, Wuppertal